CLINICAL TRIAL: NCT07216924
Title: Remapping Text in Sentence and Word Tasks to Aid Reading With Central Vision Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Remapping in reading tasks
Record Dates: First submitted 2025-09-22; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Macular Degeneration; Central Visual Impairment
Keywords: Reading; Central Field Loss
MeSH Terms: conditions — Macular Degeneration; Blindness, Cortical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Perceptual Learning (Experimental): Participants will practice reading with remapping over many sessions on different days.
  Interventions: Behavioral: Personalised Remapping Training
- Rapid Serial Visual Presentation (Experimental): Participants will read words presented one at a time in rapid succession near fixation.
  Interventions: Behavioral: RSVP personalized remappi
- Reading in The Wild (Experimental): Participants will view scenes in virtual reality showing natural settings and read a single word at a time within those scenes- e.g. a name on a street sign or shop in a city scene.
  Interventions: Behavioral: Reading text in the wild with remapping

INTERVENTIONS:
Behavioral: Personalised Remapping Training — Participants will receive training across multiple days with text being shifted in real time as it is being read from locations covered by scotoma to locations determined by personalization procedure .
  Arms: Perceptual Learning
Behavioral: RSVP personalized remappi — Participants will read one word at a time presented in rapid succession at fixation with text being shifted from scotoma locations to locations determined by personalization procedure.
  Arms: Rapid Serial Visual Presentation
Behavioral: Reading text in the wild with remapping — Participants will read short texts presented in natural scenes in virtual reality with text being shifted from scotoma locations to locations determined by personalization procedure.
  Arms: Reading in The Wild

SUMMARY:
Reading performance in patients with Central Vision Loss will be measured with and without missing text being remapped to different parts of the visual field in a variety of different reading tasks.

DETAILED DESCRIPTION:
Following initial characterization of their visual field loss, the participant's performance in various reading tasks will be measured with and without remapping. Tasks will include reading simple sentences, reading popular fiction, reading text with one word presented at a time (rapid serial visual presentation, RSVP), and reading text in simulated real-world environments in virtual reality (e.g. subway station, school, city street). Different remapping strategies, e.g. mainly shifting the text horizontally, or vertically, will be tested.

Participants interested in the study will be brought in for an initial visit where they will first be consented. Participants will then undergo a standard exam at the UMN eye clinic, if they have not had one within the last month. Participants will then have their scotomas mapped using a microperimeter housed in the Ophthalmology department to give size and shape information. Participants will perform visual tasks that are used as the basis of their personalized remapping, letter perimetry. Participants will first view and report three randomly selected horizontally arranged letters placed at different locations in the visual field. This letter perimetry task will take about 40 min and will cover a large part of the visual field. Participants will then read single words whose letters have been displaced from horizontal in various ways that comprise candidate remappings generated on the basis of the letter perimetry results. This personalization test will take about 40 minutes, and will find a good remapping strategy for the individual. Subjects will then be introduced to the reading tasks that comprise the remainder of the study The study then branches into three arms. In one arm, participants will be given repeated practice reading sentences with remappings. In XX additional sessions, participants will perform a single sentence reading tasks for remapped and non-remapped text: One sentence at a time will be displayed on the screen, and the task is simply to read aloud what was presented. Following blocks of this task with and without remapping, participants will be given extended practice reading with remapping. Participants read multiple sentences from a longer text (popular fiction) in multiple 10 minute blocks. Each sentence will be presented individually, and participants will continuously read one sentence after another taken from the fiction text.

In a second arm, participants will read sentences with one word at a time presented in rapid succession. This form of reading is called rapid serial visual presentation or RSVP. In an initial block of sentences, different word rates will be tested to determine the fastest rate where participants are accurate, with and without remapping. Then individual sentences and longer passages will be read as in the other arm, but with this different presentation method. Different remappings and no remapping will again be tested.

In a third arm, participants will read single words presented in naturalistic scenes viewed in a virtual reality environment and presented on a head mounted display. Words will be read with and without remapping. Several different environments will be tested (e.g. subway station, school, city street). The words will be natural text that could be found in these environments, e.g. subway station names, messages on a chalkboard, storefront shop names, etc.

In all sessions in all arms, the eye tracker will be calibrated to participants' individual head and eye position. This will involve fixating at different points on the device screen (HMD or desk-mounted) as the eye is imaged by the eye trackers. Throughout all testing, patients will be asked if they feel any discomfort, and will be able to take a break or quit testing at any point. Reading responses will be verbal and will scored for accuracy by a research assistant.

Including the initial visit, testing for any given patient is anticipated to last no more than 16 sessions over sixteen weeks. Enrolling participants, testing, and data analysis for all participants is anticipated to take five years from the date of enrollment of the first participant.

ELIGIBILITY:
Inclusion Criteria:

* Dense bilateral scotomas of at least 2 deg diameter in each eye covering the fovea
* Bivariate contour ellipse area (BCEA) of less than 10^2 is obtained in a simple fixation task

Exclusion Criteria:

* Neovascular AMD
* Any history of visual disorders other than that causing the central vision loss.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2031-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Sentence reading speed | Measured on day 35, end of the Personalised Remapping Training in the 33 participants in the Perceptual Learning arm.
  Time it took to read sentence in words per minute
Sentence reading accuracy | Measured on day 35, end of the Personalised Remapping Training in the 33 participants in the Perceptual Learning arm.
  Percentage of correctly read words in sentence
Word reading speed: RSVP | Measured on day 21, end of the RSVP Remapping intervention in the 33 participants in the Rapid Serial Visual Presentation arm.
  Time taken to read each word
Word recognition accuracy: RSVP | Measured on day 21, end of the RSVP Remapping intervention in the 33 participants in the Rapid Serial Visual Presentation arm.
  Percentage of words correctly read
Word reading speed: Reading in The Wild | Measured on day 21, end of the Reading Text in The Wild with Remapping intervention in the 33 participants in the Reading in The Wild arm.
  Time taken to read each word
Word recognition accuracy: Reading in the wild | Measured on day 21, end of the Reading Text in The Wild with Remapping intervention in the 33 participants in the Reading in The Wild arm.
  Percentage of words correctly read

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Edina, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Psychophysical (behavioral) data on reading will be gathered from 32 participants each in 3 experiments. Scotoma shape and location and location used for fixation will also be gathered for each participant. All data will be deidentified prior to storage in the repository.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available at the end of funding, or upon result publication, whichever comes first. As noted above all relevant publications will contain the DOI that points to the relevant data. The data will be stored as long as the OSF repository remains viable; if for some reason alternative storage sites are required within the next 10 years, the PI will pick from others available and transfer the data there.
Access Criteria: We will store data on the Open Science Foundation (OSF) repository, available to most people. Computer code will be mirrored there and also stored as github repositories. We will take and store separate "snapshots" corresponding to published protocols and analyses to insure accessibility of older code as projects continue to develop. OSF allows for the creation of a DOI for projects, and a project/DOI pair will be created and associated with each aim of the present proposal. The DOI will be referenced in publications and presentations associated with each project. The behavioral data will be stored in a general purpose format (e.g. csv files), but posted analysis and presentation code will make use of MATLAB. While MATLAB is commercial software, most universities have site licenses available. The analysis code may also run in Octave, an open-source alternative to MATLAB.